CLINICAL TRIAL: NCT04289753
Title: Behavioral Economics Applications to Geriatrics Leveraging EHRs R33 Trial
Acronym: BEAGLE R33
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Southern California (Other); University of California, Los Angeles (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stephen Persell, MD, MPH, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00210358; R33AG057383 (NIH)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Prostate Specific Antigen Screening; Asymptomatic Bacteriuria; Type 2 Diabetes
Keywords: Geriatrics; Quality of care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Cluster-randomized by primary care clinic using a constrained randomization process.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief clinician education (Active Comparator): Clinicians attributed to clinics in the brief clinician education arm will receive invitation to view an online educational module and be recruited to complete an online survey at baseline and 18 months.
  Interventions: Behavioral: Brief clinician education
- Clinical decision support nudges and brief clinician education (Experimental): Clinicians attributed to clinics randomized to the clinical decision support nudges and brief clinician decision support arm will receive clinical decision support within the EHR when conditions meet alert triggering criteria. These clinicians will also receive invitation to view an online educational module and be recruited to complete an online survey at baseline and 18 months.
  Interventions: Behavioral: EHR clinical decision support nudges; Behavioral: Brief clinician education

INTERVENTIONS:
Behavioral: EHR clinical decision support nudges — Clinical decision support nudges delivered within the EHR when conditions meet alert triggering criteria.
  Arms: Clinical decision support nudges and brief clinician education
Behavioral: Brief clinician education — Clinicians will be invited to view brief education material.

SUMMARY:
Investigators will evaluate clinical decision support nudges informed by behavioral science and directed at primary care clinicians. These will be used to reduce commonly misused, and potentially harmful, diagnostic and therapeutic actions that occur in the care of older adults (e.g. overtreatment of type 2 diabetes, misuse of PSA screening, misuse of urine testing in women with nonspecific symptoms or no symptoms.

DETAILED DESCRIPTION:
Diagnostic and therapeutic strategies misapplied to older adults can lead to increased morbidity and mortality. Despite recommendations from the American Geriatrics Society for the Choosing Wisely Initiative, there are clear examples where clinicians do not often follow best practices leading to patient harm. These include: (1) testing and treatment for asymptomatic bacteriuria (ASB) in older women, (2) prostate specific antigen (PSA) screening in older men, and (3) aggressive treatment with insulin or oral hypoglycemics for type 2 diabetes.

Clinical decision support nudges, informed by behavioral economics and social psychology and delivered via electronic health records (EHRs), are promising strategies to reduce the misuse of services. Behavioral economics-informed interventions influence conscious and unconscious drivers of decision making, are low cost, and can be incorporated into existing systems.

This randomized controlled trial will evaluate the effects of three clinical decision support nudges on three clinical quality measures, indicators of patient safety, and clinician attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Northwestern Medicine primary care clinician who sees patients under department code of a randomized clinic

Exclusion Criteria:

* Resident physicians will be excluded
* Clinicians who participated in pilot study of these interventions
* Clinician study investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37134 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Persell, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Derived] Persell SD, Petito LC, Lee JY, Meeker D, Doctor JN, Goldstein NJ, Fox CR, Rowe TA, Linder JA, Chmiel R, Peprah YA, Brown T. Reducing Care Overuse in Older Patients Using Professional Norms and Accountability : A Cluster Randomized Controlled Trial. Ann Intern Med. 2024 Mar;177(3):324-334. doi: 10.7326/M23-2183. Epub 2024 Feb 6. PMID 38315997

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinic
Period: Overall Study
Arm/Group | Brief Clinician Education | Clinical Decision Support Nudges and Brief Clinician Education
Started | 18709; 30 Clinic | 18425; 30 Clinic
Completed | 18709; 30 Clinic | 18425; 30 Clinic
Not Completed | 0; 0 Clinic | 0; 0 Clinic

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Clinician Education | Clinical Decision Support Nudges and Brief Clinician Education | Total
Number analyzed (Participants) | 18709 | 18425 | 37134
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (7.5) | 77.7 (7.4) | 77.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11244 | 11435 | 22679
  Male | 7465 | 6990 | 14455
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 699 | 974 | 1673
  Non-Hispanic White | 15209 | 14721 | 29930
  Non-Hispanic Black | 1227 | 1338 | 2565
  Other | 1574 | 1392 | 2966
Region of Enrollment [Number; unit: participants]
  United States | 18709 | 18425 | 37134

OUTCOME MEASURES:

1. Primary Outcome: PSA Screening in Older Men
Description: Measure defined as the presence of a PSA laboratory result in the EHR during the measurement period among men aged 76 years and older at the start of the measurement period with at least one visit during the measurement period with a primary care clinician and who are without a diagnosis or procedure suggesting a history of prostate cancer.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Clinician Education | Clinical Decision Support Nudges and Brief Clinician Education
Number analyzed (Participants) | 5169 | 4811
Participants | 1675 | 1373
Statistical Analysis 1: Comparison: Brief Clinician Education vs Clinical Decision Support Nudges and Brief Clinician Education; Test type: Superiority; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.46 to 0.69]

2. Primary Outcome: Urine Testing for Non-specific Reasons
Description: Measure defined as the absence of a diagnostic code for a specific genitourinary sign, symptoms or other potentially relevant indication among instances where a urinalysis and/or urine culture is obtained in the interval 24 hours before to 48 hours after a face-to-face ambulatory care visit by a woman aged 65 years or older with a primary care clinician during the measurement period.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Clinician Education | Clinical Decision Support Nudges and Brief Clinician Education
Number analyzed (Participants) | 4535 | 4264
Participants | 1127 | 1032
Statistical Analysis 1: Comparison: Brief Clinician Education vs Clinical Decision Support Nudges and Brief Clinician Education; Test type: Superiority; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.55 to 0.85]

3. Primary Outcome: Diabetes Overtreatment in the Elderly
Description: Measure defined as having the most recent hemoglobin A1C during the measurement period of less than 7.0 and insulin or an oral hypoglycemic drug on their active medication list at the end of the measurement period among adults aged 75 years and older with a diagnosis of diabetes mellitus.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Clinician Education | Clinical Decision Support Nudges and Brief Clinician Education
Number analyzed (Participants) | 3781 | 3624
Participants | 603 | 605
Statistical Analysis 1: Comparison: Brief Clinician Education vs Clinical Decision Support Nudges and Brief Clinician Education; Test type: Superiority; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.70 to 1.0]

4. Secondary Outcome: Rate of UTI Requiring Hospital Care Among Women 65 and Over Following Clinical Decision Support Exposure
Description: Emergency department visit or hospitalization for an infection originating from the urinary tract within 28 days of any primary care office visit with decision support exposure.
Time Frame: 18 months
Reporting Status: Not Posted

5. Secondary Outcome: Rate of UTI Requiring Hospital Care Among Women 65 and Over Following an Office Visit
Description: Emergency department visit or hospitalization for an infection originating from the urinary tract within 28 days of any primary care office visit
Time Frame: 18 months
Reporting Status: Not Posted

6. Secondary Outcome: Rate of Hyperglycemia Requiring Hospital Care Following Clinical Decision Support Exposure
Description: Emergency department visit or hospitalization for hyperglycemia within 90 days of an index visit where the clinician was exposed to the diabetes decision support.
Time Frame: 18 months
Reporting Status: Not Posted

7. Secondary Outcome: Rate of Hyperglycemia Requiring Hospital Care Among Previously Tightly Controlled
Description: Emergency department visit or hospitalization for hyperglycemia among patients who previously had a HbA1c <7.0 and met the criteria for treatment deintensification intervention and had one or more outpatient primary care encounters during the study period.
Time Frame: 18 months
Reporting Status: Not Posted

8. Secondary Outcome: Rate of Poor Diabetes Control Among Previously Tightly Controlled
Description: Occurrence of HbA1c >9.0 among patients who previously had a HbA1c <7.0 and met the criteria for treatment deintensification intervention and had one or more outpatient primary care encounters during the study period.
Time Frame: 18 months
Reporting Status: Not Posted

9. Secondary Outcome: Rate of Hypoglycemia Requiring Urgent Care Among Previously Tightly Controlled
Description: Emergency department visit or hospitalization for hypoglycemia among patients who previously had a HbA1c <7.0 and met the criteria for treatment deintensification intervention and had one or more outpatient primary care encounters during the study period
Time Frame: 18 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: PSA Screening in Older Men
Description: as for outcome 1
Time Frame: 19-30 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Urine Testing for Non-specific Reasons
Description: as for outcome 2
Time Frame: 19-30 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Diabetes Overtreatment in the Elderly
Description: as for outcome 3
Time Frame: 19-30 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Rates of Prostate Biopsy
Description: Rate of prostate biopsy among men >=76 with at least one visit during the measurement period with a primary care clinician and who are without a diagnosis or procedure suggesting a history of prostate cancer at the beginning of the measurement period
Time Frame: 18 months and 19-30 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Rate of Prostate MRI
Description: Rate of prostate MRI among men >=76 with at least one visit during the measurement period with a primary care clinician and who are without a diagnosis or procedure suggesting a history of prostate cancer at the beginning of the measurement period
Time Frame: 18 months and 19-30 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Rate of Prostate Cancer Diagnosis
Description: Rate of prostate cancer diagnosis among men >=76 with at least one visit during the measurement period with a primary care clinician and who are without a diagnosis or procedure suggesting a history of prostate cancer at the beginning of the measurement period
Time Frame: 18 months and 19-30 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: PSA Screening Done by Non PCP in Men Over 76 Years Old
Description: Presence of a PSA laboratory result in the EHR during the measurement period among men aged 76 years and older at the start of the measurement period ordered by a non-primary care clinician and who are without a diagnosis or procedure suggesting a history of prostate cancer.
Time Frame: 18 months and 19-30 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: PSA Screening in Men Aged 55 to 69 and Age 70 to 75
Description: Measure defined as the presence of a PSA laboratory result in the EHR during the measurement period for men aged 55-69 and men aged 70-75 who are without a diagnosis suggesting a history of prostate cancer
Time Frame: 18 months and 19-30 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Rates of Urinalysis and Urine Culture Use in Women 65 and Older
Description: Proportion of all women with one or more visit to an eligible clinic during the prior 12 months receiving urinalysis and/or urine culture
Time Frame: 18 months and 19-30 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Rate of Treatment for Antibiotics for UTI in Women 65 and Older
Description: Proportion of all women with one or more encounter to an eligible clinic during the prior 12 months receiving an antibiotic for confirmed or possible UTI.
Time Frame: 18 months and 19-30 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Dose Reduction in Insulin, Sulfonylurea or Meglitinides
Description: Proportion of patients 75 years old and older with initial HbA1c <7.0 and treated with insulin, sulfonylurea or meglitinides who have a dose reduction
Time Frame: 18 months, 24 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: PSA Screening in Older Men by Race
Description: NIH-required analysis. Measure defined as the presence of a PSA laboratory result in the EHR during the measurement period among men aged 76 years and older at the start of the measurement period with at least one visit during the measurement period with a primary care clinician and who are without a diagnosis or procedure suggesting a history of prostate cancer.
Time Frame: 18 months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: PSA Screening in Older Men by Ethnicity
Description: as for outcome 21
Time Frame: 18 months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Urine Testing for Non-specific Reasons by Race
Description: NIH-required analysis. Measure defined as the absence of a diagnostic code for a specific genitourinary sign, symptoms or other potentially relevant indication among instances where a urinalysis and/or urine culture is obtained in the interval 24 hours before to 48 hours after a face-to-face ambulatory care visit by a woman aged 65 years or older with a primary care clinician during the measurement period.
Time Frame: 18 months
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Urine Testing for Non-specific Reasons by Ethnicity
Description: as for outcome 23
Time Frame: 18 months
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Diabetes Overtreatment in the Elderly by Sex
Description: NIH-required analysis. Measure defined as having the most recent hemoglobin A1C during the measurement period of less than 7.0 and insulin or an oral hypoglycemic drug on their active medication list at the end of the measurement period among adults aged 75 years and older with a diagnosis of diabetes mellitus.
Time Frame: 18 months
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Diabetes Overtreatment in the Elderly by Race
Description: as for outcome 25
Time Frame: 18 months
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Diabetes Overtreatment in the Elderly by Ethnicity
Description: as for outcome 25
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: These adverse event data were collected over 18-month trial intervention period.
Description: All adverse event outcomes were systematically queried for using electronic health record data.
  Each adverse event is for a specific, separate clinical outcome. The denominators of patients 'at risk' differ by adverse event. For example, male patients who were included in denominator for diabetes outcomes are not 'at risk' for interventions or outcome denominators aimed at urine studies for female patients.
Arm/Group | Brief Clinician Education | Clinical Decision Support Nudges and Brief Clinician Education
All-Cause Mortality (participants affected / at risk) | 511/18709 | 469/18425
Serious Adverse Events (participants affected / at risk) | 996/38607 | 1100/35786
Other Adverse Events (participants affected / at risk) | 11/668 | 22/782
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brief Clinician Education (N=38607) | Clinical Decision Support Nudges and Brief Clinician Education (N=35786)
EHR-identified ED or hospital care possibly due to UTI or sepsis (Renal and urinary disorders) | 977 | 1090 — EHR-identified ED or hospital care possibly due to UTI or sepsis among women 65 and over following an office visit. Adverse event were assessed for the specific population of subjects to which this measure applies.
EHR-Identified ED or hospital care possibly due to hyperglycemia (General disorders) | 19 | 10 — EHR-Identified ED or hospital care possibly due to hyperglycemia among previously tightly controlled. Adverse event were assessed for the specific population of subjects to which this measure applies.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brief Clinician Education (N=668) | Clinical Decision Support Nudges and Brief Clinician Education (N=782)
Poor diabetes control (General disorders) | 11 | 22 — Poor diabetes control among previously tightly controlled. Adverse event were assessed for the specific population of subjects to which this measure applies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT04289753/Prot_SAP_000.pdf